CLINICAL TRIAL: NCT06911866
Title: A Phase Ib Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, Immunogenicity and Preliminary Efficacy of RC1416 Injection in Patients With Moderate to Severe Asthma
Brief Title: A Phase Ib Study of RC1416 Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing RegeneCore Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RJK-RC1416-102
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-03

CONDITIONS: Moderate to Severe Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RC1416 (Experimental)
  Interventions: Drug: RC1416
- Placebo (Placebo Comparator)
  Interventions: Drug: RC1416 Placebo

INTERVENTIONS:
Drug: RC1416 — there are four doses(200mg-400mg) in this part. Each subjects will receive the drug once by subcutaneous injection.
  Arms: RC1416
Drug: RC1416 Placebo — Each subjects will receive the placebo once by subcutaneous injection.
  Arms: Placebo

SUMMARY:
This is a Phase Ib study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, immunogenicity and preliminary efficacy of RC1416 injection in patients with moderate to severe asthma.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled, ascending dose Phase Ib clinical study. RC1416 is a bispecific antibodies .It is being developed by Nanjing RegeneCore Biotech Co., Ltd. as a potential therapy for asthma. A total 40 patients with moderate to severe asthma will be enrolled in 4 groups to access the safety, tolerability, PK, PD, immunogenicity and preliminary efficacy of RC1416 injection.

ELIGIBILITY:
Inclusion Criteria:

1. The subject fully understands the purpose, nature, methods and potential adverse events of the trial and voluntarily signs the informed consent form (ICF);
2. Male or female patients aged ≥18 and ≤75 years at the time of ICF signing;
3. The subject has been diagnosed with asthma for at least one year;
4. The subject has been treated with medium to high-dose inhaled corticosteroids (ICS) (e.g.,fluticasone propionate ≥ 250 μg daily or equivalent ICS dose) in combination with at least one additional controller medication [such as long-acting β2 receptor agonists (LABA), long-acting anticholinergic drugs (LAMA), leukotriene receptor antagonists (LTRA), or sustained-release theophylline] for ≥ 3 months prior to ICF signing, with a stable dosing for ≥ 1 month before randomization;
5. ACQ-6 score > 1.5 or ACT score < 20 ;
6. Pre-bronchodilator FEV1 ≤ 80% of predicted value at screening;
7. Positive objective tests for variable airflow obstruction within one year before randomization or during the screening period (including bronchodilation test, bronchial provocation test or peak expiratory flow variability, etc.).
8. The subject agrees to take effective contraceptive measures (as specified in the protocol) from the time of ICF signing until 6 months post-treatment.

Exclusion Criteria:

1. Based on the investigator's judgment,Clinically diagnosed with chronic obstructive pulmonary disease (COPD) or other lung diseases that may significantly impair lung function (such as atelectasis, pulmonary fibrosis, bronchopulmonary dysplasia, bronchiectasis, emphysema, etc.) ;
2. Subjects who had required at least one systemic glucocorticoid treatment due to asthma exacerbation or other reasons, or who had been hospitalized or treated emergency department due to asthma exacerbation within one month before administration;
3. Subjects with a history of near-fatal asthma requiring endotracheal intubation and mechanical ventilation;
4. Subjects who are Excessive dependence on short-acting β-agonists (SABA) (>10-12 puffs per day) , especially use more than one vial of salbutamol (or equivalent) per month;
5. Subjects who used non-selective β-blockers within 1 month before screening until randomization;
6. Subjects with pulmonary or other infection and oral or intravenous antibiotics or antifungal or antiviral drugs within one month before administration; Subjects have need local antibiotic or antiviral treatment within 7 days before screening;Subjects with a history of recurrent infections (≥3 times per year) and underlying diseases that predispose to infection; Subjects with a history of disseminated herpes simplex infection or recurrent (>1 time) or disseminated herpes zoster; Subjects with a history of opportunistic infections;
7. Subjects who underwent major surgery within 6 months prior to screening or planned major surgery during the trial.
8. Subjects who have suffered form malignancy within 5 years,except:

   * Subjects with cervical carcinoma in situ that has been completely resected and has no evidence of recurrence or metastasis for at least 3 years;
   * Subjects with basal cell or squamous cell carcinoma that have been completely resected and have no recurrence for at least 3 years;
   * Subjects with a history of cancer who have had complete remission of their malignant tumors for at least 5 years at the time of screening and have no anti-tumor treatment;
9. Currently receiving or having received any of the prohibited drugs or treatments in this trial within the following time frames :

   1. Live vaccines, attenuated live vaccines, or adenovirus vector vaccines within 3 months prior to screening or plan to receive such vaccines during the trial;
   2. Any of the following drugs within 3 months or 5 half-lives (whichever is longer) prior to screening: IL-4Rα antagonists, IL-5/interleukin-5 receptor (IL-5R) antagonists, anti-IgE monoclonal antibodies, anti-TSLP antibodies, etc.;
   3. Bronchial thermoplasty within 3 years prior to screening;
   4. Allergen immunotherapy within 3 months prior to screening or plan to receive such treatments during the trial;
   5. Drugs that affect immunity within 3 months or 5 half-lives (whichever is longer) prior to screening, including but not limited to systemic immunosuppressants/immunomodulatory drugs (including but not limited to methotrexate, cyclosporine, etc.);
   6. Montelukast within 2 weeks prior to screening;
   7. Immunoglobulin products within 3 months prior to screening;
   8. Traditional Chinese medicine or herbal products that affect bronchospasm and/or lung function within 1 month prior to screening.
10. Subjects who have received any investigational drug or participated in other clinical trials or medical research activities within 3 months or 5 half-lives (whichever is longer) before screening, or plan to participate in other drug or medical device clinical trials during the trial; except subjects who have only signed the ICF and participated in the screening of clinical trials but did not receive clinical trial treatment or enrollment within 3 months before the first dose.
11. Subjects who have donated blood or lost blood ≥ 400 mL (excluding menstrual blood loss), or received blood transfusion or used blood products within 3 months before screening, or plan to donate blood during the study or within 1 month after the end of the trial.
12. Current smokers or subjects who quit smoking within 6 months before screening, or previous smokers who quit smoking more than 6 months at screening with a smoking history > 10 pack-years (pack-years = number of packs smoked per day × number of years of smoking, 20 cigarettes per pack), or who cannot quit smoking during the trial.
13. Subjects with known to be allergy to the excipients or ingredients of this product, or have had severe drug or food allergic reactions in the past.
14. With any psychological disorders or neurological/psychiatric disorders confirmed by the investigator.
15. Subjects who have difficulty with venous blood collection,or are afraid of needles or blood, or those who have difficulty with subcutaneous injection administration.
16. Any of the following abnormal in laboratory test results at screening or baseline:

    1. Hemoglobin < 90 g/L;
    2. Platelet count < 100 × 109/L;
    3. Absolute neutrophil count (ANC) < 1.2 × 109/L;
    4. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 × ULN (upper limit of normal);
    5. Serum creatinine > 1.5 × ULN;
    6. Total bilirubin > 1.5 × ULN;
    7. Other laboratory test results abnormalities are clinically significant, and the investigator judge that the subject are unsuitable for enrollment.
17. Subject with clinically significant abnormalities in the 12-lead ECG at screening or baseline as judged by the investigator , or prolonged QTc ( QTcF interval >450 ms for males and >470 ms for females, Corrected by Fridericia，s formula), or a history of long QT syndrome.
18. Any one of infectious disease screening indicators meets the following criteria at screening:

    1. According to the judgment of the investigator, there is vidence of active tuberculosis or a history of active tuberculosis without appropriate treatment, and screening results suggest the possibility of latent tuberculosis infection as judged by the investigator;
    2. Positive for hepatitis B surface antigen (HBsAg), or positive for hepatitis B core antibody (HBcAb) and hepatitis B virus deoxyribonucleic acid (HBV DNA) exceeds the detection limit;
    3. Hepatitis C antibody (HCVAb) positive and hepatitis C virus ribonucleic acid (HCV RNA) exceeds the detection limit;
    4. Positive for Treponema pallidum (Tp) antibody;
    5. Positive for human immunodeficiency virus antigen (HIVAg) or human immunodeficiency virus antibody (HIVAb).
19. Subject with previous history of drug abuse/drug use；
20. Subject with a history of alcoholism within 6 months prior to screening[(i.e., more than 14 standard units per week for women and more than 21 standard units per week for men (1 standard unit containing 14g of alcohol, such as 360 mL beer or 45 mL spirits with 40% alcohol or 150 mL wine) ]or those who cannot abstinence during the trial;
21. Pregnant or lactating women, or those with a positive pregnancy test result;
22. Other situations that the investigator judged are unsuitable for participating in this trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-10-25 (Actual); Primary Completion 2025-09-25 (Actual); Study Completion 2025-09-25 (Actual)

PRIMARY OUTCOMES:
AE | up to 141 days
  incidence ,severity and relation to investigational drugs of Adverse Events according to CTCAE V5.0
SAE | up to 141 days
  incidence ,severity and relation to investigational drugs of Adverse Events according to CTCAE V5.0
Vital Signs | up to 141 days
  number of praticipants with clinically notable Vital Signs according to CTCAE V5.0
Laboratory Tests | up to 141 days
  number of praticipants with clinically Laboratory Tests Values according to CTCAE V5.0
ECG | up to 141 days
  number of praticipants with clinically notable Electrocardiogram(ECG) Values according to CTCAE V5.0
Injection Site Reaction | up to 85 days
  number of praticipants with clinically notable Injection Site Reaction according to CTCAE V5.0

SECONDARY OUTCOMES:
Cmax | up to 141 days
  maximum serum concentration
AUC0-t | up to 141 days
  AUC extrapolated to infinitymeasurable concentration
AUC0-inf | up to 141 days
  area under the concentration-time curve (AUC) from administration to the last measurable concentration
Anti-Drug antibody (ADA) | up to 141 days
  number and percentage of subjects tested ADA positive
Tmax | up to 141 days
  time to reach maximum concentration
t1/2 | up to 141 days
  the terminal elimination half-life
MRT | up to 141 days
  mean residence time
λz | up to 141 days
  elimination rate constant
CL/F | up to 141 days
  apparent clearance
Vz/F | up to 141 days
  apparent volume of distribution
Change from baseline in fractional exhaled nitric oxide (FeNO) | up to 141 days
  Preliminary effectiveness indicators
Change from baseline in total IgE (immunoglobulin E), human thymus and activation-regulated chemokine (TARC) | up to 141 days
  Preliminary effectiveness indicators
Change from baseline in blood eosinophil (EOS) count, free or bound IL-5 and total IL-5, and free IL-4 and IL-13 levels | up to 141 days
  Preliminary effectiveness indicators

CONTACTS AND LOCATIONS:
Locations (16):
- China (16):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Peking University Shougang Hospital, Beijing, Beijing Municipality
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - The First Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - Hebei Petro China Centre Hospital, Langfang, Hebei
  - Hebei Province Hospital of Chinese Medicine, Shijiazhuang, Hebei
  - Nanyang Central Hospital, Nanyang, Henan
  - Xinxiang First People's Hospital, Xinxiang, Henan
  - The First Affiliated Hospital of Baotou Medical College, Baotou, Inner Mongolia
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Jining NO.1 people's hospital, Jining, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Zibo Municipal Hospital, Zibo, Shandong
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No